CLINICAL TRIAL: NCT03595085
Title: Safety and Efficacy of Catheter Directed Interventions in Acute High Risk Pulmonary Embolism
Brief Title: Catheter Directed Interventions in Pulmonary Embolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, heba ahmed hamed, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTPE
Record Dates: First submitted 2018-07-12; First posted 2018-07-23 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Fibrinolytic Agents; Streptokinase

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- catheter directed interventions (Experimental): Those patients will undergo catheter directed fragmentation followed by local thrombolysis using streptokinase
  Interventions: Procedure: catheter directed fragmentation and thrombolysis
- systemic thrombolysis (Active Comparator): Those patients will receive systemic streptokinase
  Interventions: Drug: Streptokinase

INTERVENTIONS:
Procedure: catheter directed fragmentation and thrombolysis — A(6)F multipurpose catheter will be advanced over a guide wire under fluoroscopic guidance and used to measure right heart and pulmonary artery pressures, then mechanical catheter fragmentation will be done using a pigtail catheter. The catheter will be quickly spun manually so as to fragment the central thrombus and establish initial flow into pulmonary artery. After ensuring initial flow, Initial bolus dose of streptokinase (250.000 international unit) will be given over 10 min followed by continuous infusion of (100.000 international unit per hour)for 24 hours
  Arms: catheter directed interventions
Drug: Streptokinase — intravenous streptokinase at a dose of 250 000 international unit as a loading dose over 30 minutes, followed by 100 000 international unit per hour over 12-24 hours
  Arms: systemic thrombolysis

SUMMARY:
Evaluating the safety and outcomes of catheter directed thrombolysis following catheter fragmentation in acute high risk pulmonary embolism

DETAILED DESCRIPTION:
Acute pulmonary embolism is common, but its presentation highly varies ranging from asymptomatic to massive pulmonary embolism. Massive pulmonary embolism is a common life-threatening condition and represents the most serious manifestation among venous thromboembolic disease.

Acute pulmonary embolism is considered the third most common cause of death among hospitalized patients . The mortality rate can exceed 58% in patients with acute pulmonary embolism presenting with haemodynamic instability , mostly occur within 1 hour of presentation.

In patients with high risk pulmonary embolism , the main aim of therapy is to rapidly recanalize the affected pulmonary arteries with thrombolysis or embolectomy; to decrease right ventricular afterload and reverse right ventricular failure and shock, prevent chronic thromboembolic pulmonary hypertension , and decrease the recurrence risk.

The first-line treatment in patients with acute high risk pulmonary embolism presenting with persistent hypotension and/or cardiogenic shock is intravenous thrombolytic therapy. However a significant proportion of patients may not be a candidate for Intravenous thrombolysis because of major contraindications. An alternative option in patients with absolute contraindications or has failed intravenous thrombolysis is surgical embolectomy , but the number of experienced tertiary care centers that can do emergency surgical embolectomy are limited.

Percutaneous catheter mechanical fragmentation of proximal pulmonary arterial clots followed by local thrombolytic therapy is accepted as an alternative to intravenous thrombolytic therapy and surgical embolectomy because of their ability to rapidly recanalize occluded pulmonary blood flow. Several reports have shown that catheter-directed therapy is a safe and effective treatment for acute PE to restore pulmonary flow and decreasing Pulmonary artery systolic pressure , However, current knowledge on efficacy and safety of catheter-directed therapy in management of intermediate high risk pulmonary embolism is limited.

ELIGIBILITY:
Inclusion Criteria:

* Patients with angiographically confirmed acute high risk pulmonary embolism with shock index >1.
* Pulmonary arterial occlusion with >50% involvement of the central (main and/or lobar) pulmonary , and pulmonary hypertension (mean pulmonary artery pressure >25 mmHg)
* Patients with high risk pulmonary embolism who remain unstable after receiving fibrinolysis
* Patients with high risk pulmonary embolism who cannot receive fibrinolysis
* Patients with acute intermediate-high risk pulmonary embolism with adverse prognosis (new hemodynamic instability, worsening respiratory failure, severe RV dysfunction, or major myocardial necrosis)

Exclusion Criteria:

* Patients with echocardiographically confirmed right sided thrombi.
* Patients with low-risk pulmonary embolism or intermediater-low risk acute pulmonary embolism with minor RV dysfunction, minor myocardial necrosis, and no clinical worsening
* Acute gastrointestinal bleeding.
* Anticoagulation with international normalized ratio >1.8 or severe coagulopathy.
* Anaphylactic reaction to contrast media.
* Acute stroke.
* Acute renal failure or severe chronic non-dialysis dependent kidney disease.
* Uncooperative patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  measure the estimates of deaths in the 30 days after pulmonary embolism diagnosis

SECONDARY OUTCOMES:
Changes in blood pressure | 24 hours
  systolic and diastolic blood pressure will be measured at first admission and compared with measurements the following second, eighth, and 24th hours of the intervention
oxygen saturation | 24 hours
  oxygen saturation will be measured by arterial blood gases analysis at first admission and compared with measurements the following second, eighth, and 24th hours of the intervention
changes in right ventricular dysfunction | 24 hours
  right ventricular dysfunction will be assessed by echocardiography and Mean pulmonary artery systolic pressure will be estimated by transthoracic echocardiography at first admission and 24 hours after catheter-directed intervention

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heit JA. The epidemiology of venous thromboembolism in the community. Arterioscler Thromb Vasc Biol. 2008 Mar;28(3):370-2. doi: 10.1161/ATVBAHA.108.162545. No abstract available. PMID 18296591
- [Background] Konstantinides SV, Torbicki A, Agnelli G, Danchin N, Fitzmaurice D, Galie N, Gibbs JS, Huisman MV, Humbert M, Kucher N, Lang I, Lankeit M, Lekakis J, Maack C, Mayer E, Meneveau N, Perrier A, Pruszczyk P, Rasmussen LH, Schindler TH, Svitil P, Vonk Noordegraaf A, Zamorano JL, Zompatori M; Task Force for the Diagnosis and Management of Acute Pulmonary Embolism of the European Society of Cardiology (ESC). 2014 ESC guidelines on the diagnosis and management of acute pulmonary embolism. Eur Heart J. 2014 Nov 14;35(43):3033-69, 3069a-3069k. doi: 10.1093/eurheartj/ehu283. Epub 2014 Aug 29. No abstract available. PMID 25173341
- [Background] Uflacker R. Interventional therapy for pulmonary embolism. J Vasc Interv Radiol. 2001 Feb;12(2):147-64. doi: 10.1016/s1051-0443(07)61821-1. PMID 11265879
- [Background] Kasper W, Konstantinides S, Geibel A, Olschewski M, Heinrich F, Grosser KD, Rauber K, Iversen S, Redecker M, Kienast J. Management strategies and determinants of outcome in acute major pulmonary embolism: results of a multicenter registry. J Am Coll Cardiol. 1997 Nov 1;30(5):1165-71. doi: 10.1016/s0735-1097(97)00319-7. PMID 9350909
- [Background] Stein PD, Alnas M, Beemath A, Patel NR. Outcome of pulmonary embolectomy. Am J Cardiol. 2007 Feb 1;99(3):421-3. doi: 10.1016/j.amjcard.2006.08.050. Epub 2006 Dec 15. PMID 17261411
- [Background] Engelberger RP, Kucher N. Reperfusion Treatment for Acute Pulmonary Embolism. Hamostaseologie. 2018 May;38(2):98-105. doi: 10.1055/s-0038-1641717. Epub 2018 May 29. PMID 29843174
- [Background] Kuo WT, Banerjee A, Kim PS, DeMarco FJ Jr, Levy JR, Facchini FR, Unver K, Bertini MJ, Sista AK, Hall MJ, Rosenberg JK, De Gregorio MA. Pulmonary Embolism Response to Fragmentation, Embolectomy, and Catheter Thrombolysis (PERFECT): Initial Results From a Prospective Multicenter Registry. Chest. 2015 Sep;148(3):667-673. doi: 10.1378/chest.15-0119. PMID 25856269
- [Background] Mohan B, Chhabra ST, Aslam N, Wander GS, Sood NK, Verma S, Mehra AK, Sharma S. Mechanical breakdown and thrombolysis in subacute massive pulmonary embolism: A prospective trial. World J Cardiol. 2013 May 26;5(5):141-7. doi: 10.4330/wjc.v5.i5.141. PMID 23710301
- [Background] Dilektasli AG, Demirdogen Cetinoglu E, Acet NA, Erdogan C, Ursavas A, Ozkaya G, Coskun F, Karadag M, Ege E. Catheter-Directed Therapy in Acute Pulmonary Embolism with Right Ventricular Dysfunction: A Promising Modality to Provide Early Hemodynamic Recovery. Med Sci Monit. 2016 Apr 15;22:1265-73. doi: 10.12659/msm.897617. PMID 27081754